CLINICAL TRIAL: NCT03749733
Title: Single Site, Open-label, Randomized, Two Treatments, Two Periods, Two Sequences, Crossover Single-dose Trial to Investigate the Bioequivalence of Two Oral Formulations of a Fixed-dose Combination Tablet Containing 1.5 mg Estradiol and 2.5 mg Nomegestrol Acetate (Product of Laboratorios Andrómaco S.A. [Test Product] Versus Stezza, Product of Merck Sharp & Dohme Farmacêutica Ltda. [Reference Product]) in Postmenopausal Women Under Fasting Conditions
Brief Title: Bioequivalence of Two Fixed-dose Combination Tablets Containing Estradiol and Nomegestrol Acetate
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ESTNMG-04-GRU; HP8010-01 (Other: Grünenthal); 17-CI-09 012 084 (Registry Identifier: Comisión Federal para la Protección contra Riesgos Sanitarios [COFEPRIS])
Record Dates: First submitted 2018-11-09; First posted 2018-11-21 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Bioequivalence
Keywords: Bioequivalence; Estradiol; Nomegestrol acetate
MeSH Terms: interventions — Estradiol; nomegestrol acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Participants will receive a single film-coated tablet of the test formulation containing estradiol 1.5 mg/nomegestrol acetate 2.5 mg.
  The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Estradiol 1.5 mg/nomegestrol acetate 2.5 mg (Test Product)
- Reference Product (Active Comparator): Participants will receive a single film-coated tablet of the marketed reference formulation containing estradiol 1.5 mg/nomegestrol acetate 2.5 mg.
  The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Estradiol 1.5 mg/nomegestrol acetate 2.5 mg (Reference Product)

INTERVENTIONS:
Drug: Estradiol 1.5 mg/nomegestrol acetate 2.5 mg (Reference Product) — Marketed Drug
  Other Names: Stezza (Trade Mark)
  Arms: Reference Product
Drug: Estradiol 1.5 mg/nomegestrol acetate 2.5 mg (Test Product) — Investigational Medicinal Product
  Arms: Test Product

SUMMARY:
This study will investigate the bioavailability in fasting post-menopausal women of 2 film-coated tablet formulations containing 1.5 milligrams (mg) of estradiol and 2.5 mg of nomegestrol acetate.

The study will be performed at a single site. Participants will take a single oral dose of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 21 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of estradiol and nomegestrol of 2 film-coated tablet formulations with estradiol 1.5 mg and nomegestrol acetate 2.5 mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

1. Test Product: new product manufactured by Laboratorios Andrómaco S.A.
2. Reference Product: Stezza [Trademark], product of Merck Sharp & Dohme Farmacêutica Ltda.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total estradiol/estrone and nomegestrol will be determined.

Participants will be confined in the study site for approximately 36 hours during each study period (for 12 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples will be obtained. Three blood samples will be taken before the film-coated tablet is administered (at pre-dose: -1.0, -0.5, and 0 h) and 16 samples up to 24 hours after the administration in each period. Participants will return to the site to provide additional blood samples at 36 h, 48 h, and 72 h post-dose.

The washout period between the two study periods will be at least 21 days.

The samples from each participant will be analyzed with 2 methods of high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total estradiol/estrone and nomegestrol in plasma with citrate phosphate dextrose anticoagulant. The blood samples taken at pre-dose will be taken to establish the baseline concentrations of total estrone and estradiol. The baseline-corrected and uncorrected AUCs and Cmax will be calculated.

The safety objective is to evaluate the tolerability of both formulations in post-menopausal women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

A. Participation will be voluntary and according to the guidelines proposed by the Health General Law (Mexico), and informed consent will be obtained according to the previously mentioned law. In addition, the study will be conducted according to the ethical principles that have their origin in the Declaration of Helsinki, the current Brazilian laws, and Good Clinical Practice.

B. Only post-menopausal women aged between 40 years and 65 years who meet any of the following criteria:

1. 12 months of spontaneous amenorrhea.
2. 6 months of spontaneous amenorrhea with follicle-stimulating hormone levels above 40 international units per liter and below 20 nanograms per liter estradiol.
3. Bilateral oophorectomy with or without hysterectomy.

C. The body mass index must be between 18.5 and 29.99 kilograms per square meter according to the Quetelet index.

D. Participants must be healthy determined by the results of a complete clinical history recorded by the clinical investigational site physicians and the results of the laboratory examinations done by a certified clinical laboratory.

E. Participants with pre-existing illnesses must be controlled with stable doses of medication for a period of at least 3 months.

F. Non-smoker and/or not having used nicotine or nicotine-containing products (e.g., nicotine plasters) within 3 months prior to the beginning of the study.

G. The allowed limits of variation within normal in the screening visit will be: systolic blood pressure (sitting) below 120 mmHg, diastolic blood pressure below 80 mmHg, heart rate between 50 and 100 beats per minute and respiratory rate between 14 and 20 breaths per minute according to the current standard operating procedure. Vital signs will be measured after 10 minutes of resting in a sitting position.

H. Laboratory and other examinations to be conducted for the inclusion of participants will be:

1. Complete blood count: leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, erythrocyte distribution width, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
2. Blood chemistry 27 elements: glucose, urea, blood urea nitrogen (BUN), creatinine, BUN/creatinine ratio, uric acid, cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, low-density lipoprotein (LDL), cholesterol, non-HDL cholesterol, atherogenic index, total protein, albumin, globulins, albumin/globulin ratio, total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, total alkaline phosphatase, gamma-glutamyl transferase, lactate dehydrogenase, iron, calcium, sodium, potassium, and chloride.
3. Urinalysis: Physical examination (color, appearance, density); chemical examination (pH, leukocytes, nitrite, protein, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysmorphic erythrocytes, casts, crystals, squamous epithelial cells, tubular renal cells, mucus, bacteria and yeasts).
4. Hepatitis B screening (Antibody to hepatitis B core antigen [Anti-HBc], antibody to hepatitis B surface antigen [HBs-Ab], antibody to hepatitis B surface antigen [Anti-HBs]) and hepatitis C antibodies.
5. HIV test: Antibodies to the human immunodeficiency virus (Anti-HIV 1 and 2).
6. Venereal disease research laboratory test (VDRL).
7. Urine drugs of abuse test at the screening visit and on Day 0 (approximately 12 hours prior to the administration of the investigational medicinal product [IMP] on the previous day) on both study periods.
8. Alcohol breath test on Day 0 (prior to the administration of the investigational medicinal product on the previous day) on both study periods.
9. 12-lead electrocardiogram which will be performed after resting for 10 minutes in a sitting position.

In addition, each participant will undergo the following examinations:

1. Complete gynecological profile:

   * Follicle-stimulating hormone (FSH).
   * Luteinizing hormone (LH).
   * Serum estradiol.
   * Serum progesterone.
   * Serum prolactin.
2. Bilateral mammography (with Breast Imaging Reporting and Data System [BI-RADS] 1 or 2 results).
3. Transvaginal ultrasound (without clinically significant findings).
4. Pap smear (without clinically significant findings).

Exclusion Criteria:

A. Participants with a history of the following diseases: cardiovascular (myocardial infarction, not-controlled hypertension, thromboembolic arterial or venous diseases), renal (kidney failure), hepatic (hepatitis, jaundice), muscular, metabolic, gastrointestinal, neurologic (cerebrovascular disease), psychiatric (depression) endocrinological (not-controlled diabetes mellitus), hematopoietic, respiratory or other organic abnormalities that are not appropriately controlled and that require a pharmacological treatment that could result in a drug interaction with the study medication. Women who have had muscular trauma within 21 days previous to the study will also be excluded.

B. History of major surgeries (cranial surgery, thorax, abdomen or extensive surgeries in extremity requiring the use of general or regional anesthesia and/or respiratory support) within 3 months previous to the study.

C. Participants with a history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer.

D. History of lactose intolerance.

E. Participants who have been exposed to medications known to be hepatic enzyme inducers or inhibitors within 72 hours previous to the start of the study.

F. Participants who have taken any type of vitamin supplements (with or without prescription) or herbal remedies within 30 days (or 7 half-lives) previous to the start of the study.

G. Participants undergoing hormone replacement therapy or taking thyroid hormones.

H. Participants with uterine bleeding.

I. Participants with endometrial thickness equal to or greater than 7 mm as determined in the transvaginal ultrasound.

J. Participants who have been hospitalized for any reason within 6 months prior to study start.

K. Participants who have taken investigational medicinal products from other investigations within 180 days (i.e., 6 months) prior to study start.

L. Participants with a history of allergy or hypersensitivity to the study medication (estradiol/nomegestrol), any other medication, food, or substance.

M. Participants who have consumed alcohol, carbonated beverages, or beverages that contain methylxanthines (coffee, tea, cocoa, chocolate, mate, cola, etc.), grapefruit juice, or charbroiled foods within 12 hours prior to the start of the hospitalization period.

N. Participants with any of the following results for hepatitis B: acute infection, chronic infection, or unclear result based on the interpretation of results of the hepatitis B virus serology (CDC Interpretation of Hepatitis B Serologic Test Results).

O. Participants who have donated or lost more than 450 milliliters of blood within 90 days prior to study start.

P. Participants with a history of dependence/abuse of alcohol or psychoactive substances.

Q. Participants requiring a special diet for any reason e.g., vegetarian.

R. Participants unable to understand the nature, objectives, and possible consequences of the study.

S. Evidence of the participant's uncooperativeness during the conduct of the study (unable follow the instructions and requirements of the study personnel).

T. Positive results for drugs of abuse or alcohol breath tests.

U. Participants who are not registered in the Comisión Federal para la Protección contra Riesgos Sanitarios [COFEPRIS]) webpage.

V. Relationship of subordination between the participants and the investigators.

W. Sponsor or clinical site employees.

Discontinuation criteria:

A. Safety and well-being of the participant.

B. Lack of adherence to the procedures and therefore non-compliance with the protocol.

C. Medical reasons (serious adverse events), adverse reactions to the study medication classified as severe.

D. Uncooperative attitude during the conduct of the study (unable follow the instructions and requirements of the study personnel).

E. Recurring or intercurrent disease (not controlled).

F. Withdrawal of consent to participate in the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Total estrone (corrected): area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The samples taken at pre-dose will be taken to establish the baseline concentration of total estrone. The baseline-corrected AUC0-t will be calculated.
Total estradiol (corrected): area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The samples taken at pre-dose will be taken to establish the baseline concentration of total estradiol. The baseline-corrected AUC0-t will be calculated.
Total nomegestrol: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The samples taken at pre-dose will be taken to establish the baseline concentration of total nomegestrol. The AUC0-72 will be calculated.
Total estrone (corrected): Maximum plasma concentration (Cmax) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The baseline-corrected Cmax of estrone will be calculated.
Total estradiol (corrected): Maximum plasma concentration (Cmax) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The baseline-corrected Cmax of estradiol will be calculated.
Total nomegestrol: Maximum plasma concentration (Cmax) | From tablet intake up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The achieved Cmax of nomegestrol will be calculated.

SECONDARY OUTCOMES:
Total estrone: Time to achieve maximum plasma concentration (tmax) | From tablet intake up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The tmax of estrone will be calculated.
Total estradiol: Time to achieve maximum plasma concentration (tmax) | From tablet intake up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The tmax of estradiol will be calculated.
Total nomegestrol: Time to achieve maximum plasma concentration (tmax) | From tablet intake up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The tmax of nomegestrol will be calculated.
Total estrone (uncorrected): area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The samples taken at pre-dose will be taken to establish the baseline concentration of total estrone. The AUC0-t will be calculated.
Total estradiol (uncorrected): area under the plasma concentration-time curve from 0 to time t (AUC0-t) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The samples taken at pre-dose will be taken to establish the baseline concentration of total estrone. The AUC0-t will be calculated.
Total estrone (uncorrected): Maximum plasma concentration (Cmax) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The achieved Cmax of estrone will be calculated.
Total estradiol (uncorrected): Maximum plasma concentration (Cmax) | Blood samples drawn at baseline (up to 1 hour before tablet intake) and up to 72 hours after tablet intake
  Three blood samples will be taken before the medication is administered and 19 samples up to 72 hours after the administration in each period. The achieved Cmax of estradiol will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Investigacíon Farmacológica y Biofarmacéutica (IFaB), S.A.P.I. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site (see URL below for details)
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials